CLINICAL TRIAL: NCT02950311
Title: A Prospective, Randomized, Double-blinded, Placebo-controlled Pilot Study for Evaluating the Effectiveness of Intranasal Xylitol in Treating Otitis Media With Effusion (OME) in Children
Brief Title: Xylitol for Otitis Media
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: On clinical hold with the FDA. Insufficient funds to conduct the study
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00072658
Record Dates: First submitted 2016-10-19; First posted 2016-11-01 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Otitis Media With Effusion
MeSH Terms: conditions — Otitis Media with Effusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal xylitol spray (Experimental): Two sprays each nostril, twice a day.
  Interventions: Drug: Intranasal xylitol spray
- Intranasal saline spray (Placebo Comparator): Two sprays each nostril, twice a day.
  Interventions: Other: Intranasal saline spray

INTERVENTIONS:
Drug: Intranasal xylitol spray — Two sprays into each nostril of intranasal xylitol spray will be administered to pediatric patients by parent(s)/caregiver(s) twice daily for 24 weeks.
  Arms: Intranasal xylitol spray
Other: Intranasal saline spray — Two sprays into each nostril of intranasal xylitol spray will be administered to pediatric patients by parent(s)/caregiver(s) twice daily for 24 weeks.
  Other Names: Placebo spray
  Arms: Intranasal saline spray

SUMMARY:
This is a randomized, double-blind, placebo-controlled study of children, age 6 months to 3 years, with a diagnosis of Otis media with effusion (OME) based on examination by a provider at a Duke- affiliated otolaryngology clinic.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the efficacy of intranasal xylitol in young children with otitis media with effusion as measured by the resolution of middle ear effusion based on physical examination and tympanometry at 6-, 12-, and 18 and 24-weeks post-treatment. Eligible subjects will be randomly assigned to receive either intranasal xylitol spray or a nasal saline spray placebo and will be observed for 24-weeks following initiation of daily xylitol spray or placebo. The primary efficacy endpoint, the time to middle ear effusion resolution with and without the xylitol nasal spray, will be analyzed using either a two-sample t-test or non-parametric Wilcoxon test, depending on whether the time is normal or non-normal. Risks include epistaxis, diarrhea, and allergic reaction. Serious adverse events are not anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Between 6 months and 3 years of age.
* Clinical diagnosis of OME. Treated at Duke for the above condition.
* Ability of parent/guardian to be compliant with at-home nasal spray administration.

Exclusion Criteria:

* History of immunodeficiency or an immunologic disorder that predisposes to frequent infections.
* History of prior pressure-equalization (PE) tube placement and the tubes are still in place.
* Active or recent (<1 month prior to screening) middle ear disease, including but not limited to: cholesteatoma, tympanic membrane perforation, congenital external or middle ear abnormalities or malformations.
* History of previous otologic surgery including tympanoplasty, and/or mastoidectomy.
* Previous use of intranasal sprays other than normal saline, including intranasal steroids, and/or xylitol within 1 month prior to screening.
* Any other clinically significant illness or medical condition, per PI discretion, that would prohibit the subject from participating in the study.
* Subject has previously been randomized to a trial of Xylitol.
* Parent/guardian is unable to administer the study nasal spray.
* Parent/guardian is unable to read, write, and understand English.
* Parent/guardian is unable to provide legally effective consent.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Time to middle ear effusion resolution | 24 weeks

SECONDARY OUTCOMES:
To evaluate the effect of intranasal xylitol on resolution of the conductive hearing loss associated with middle ear effusion | 24 weeks
  Results from both audiometry and tympanometry testing are combined to have a comprehensive assessment of conductive hearing loss.
Effect of intranasal xylitol on frequency of episodes of acute otitis media and sinonasal symptoms | 24 weeks
Tolerability and side effects of intranasal xylitol administration in children | 24 weeks
  Will be evaluated descriptively and include all subjects exposed to at least one dose of study drug
Tympanostomy tube (TT) placement need | 24 weeks
  The number of subjects that need TT placement in each arm will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Ryan, MD, Principal Investigator — Duke University